CLINICAL TRIAL: NCT05629234
Title: ROSY-T: Roll Over StudY for Patients Who Have Completed a Previous Oncology Study With Osimertinib and Are Judged by the Investigator to Clinically Benefit From Continued Treatment
Brief Title: Roll Over StudY for Patients Who Have Completed a Previous Oncology Study With Osimertinib (TAGRISSO) (ROSY-T)
Acronym: ROSY-T
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D5161N00007
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Cancer; Oncology; Clinically Benefit; Roll Over StudY
MeSH Terms: conditions — Neoplasms | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Osimertinib (Experimental): Participants will receive Osimertinib
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib (dose range of 40 mg to 240 mg orally, once daily)
  Other Names: TAGRISSO

SUMMARY:
The rationale of the ROSY-T study is to continue to provide study treatment for patients who have participated in a parent study with osimertinib and who are continuing to derive clinical benefit from treatment at the end of such studies, as judged by the Investigator.

DETAILED DESCRIPTION:
ROSY-T is an open label, non-randomised, multicentre, international trial for patients who have completed a parent study using osimertinib and who are deriving clinical benefit from continued treatment as judged by the Investigator. Patients will be rolled-over from the parent study and will continue the study, until they meet one of the treatment discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written Informed Consent Form (ICF).
2. Patient is currently deriving clinical benefit from continued treatment with osimertinib in an AstraZeneca parent study using osimertinib monotherapy which has met its endpoints or has otherwise stopped.
3. Patients should be using adequate contraceptive measures.

Exclusion Criteria:

1. Ongoing, unresolved, Grade 3 or above toxicity requiring interruption of treatment at the time of the termination of the parent study.
2. Currently receiving treatment with any prohibited medication(s).
3. Concurrently enrolled in any other type of medical research judged not to be scientifically, or medically compatible with this study.
4. Permanent discontinuation from the parent study due to toxicity or disease progression.
5. Local access to commercially-available drug at no cost to the patient is permitted by local regulation.

Exclusion Criteria for the sub-study:

1. Active infection including active hepatitis C and Human immunodeficiency virus (HIV) infection or active uncontrolled Hepatitis B virus (HBV) infection. Screening for chronic conditions is not required.

Patients with HBV infection are only eligible if they meet all the following criteria:

* Demonstrated absence of HCV co-infection or history of HCV co-infection;
* Demonstrated absence of HIV infection;
* Patients receiving anti-viral treatment for at least 6 weeks prior to study treatment, HBV DNA is suppressed to < 100 IU/mL, and transaminase levels are below ULN.

Patients with a resolved or chronic HBV infection are eligible if they are:

* Negative for HBsAg and positive for anti-HBc IgG. In addition, patients must be receiving anti-viral prophylaxis for 2 to 4 weeks prior to study treatment and 6 to 12 months (to be determined by hepatologist) post treatment; or
* Positive for HBsAg, but for > 6 months have had transaminases levels below ULN and HBV DNA levels below < 100 IU/mL (ie, patients are in an inactive carrier state). In addition, patients must be receiving anti-viral prophylaxis for 2 to 4 weeks prior to study treatment.

Should participants with HIV infection be included, patients are only eligible if they meet all the following criteria:

* Undetectable viral RNA load for 6 months
* CD4+ count of > 350 cells/μL
* No history of AIDS-defining opportunistic infection within the past 12 months (to be determined by hepatologist) post treatment
* Stable for at least 4 weeks on anti-HIV medications.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) | Until 90 days after the last dose of study treatment
  Safety and tolerability of osimertinib will be assessed.

CONTACTS AND LOCATIONS:
Locations (21):
- China (4):
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- Research Site, Villejuif, France
- Malaysia (4):
  - Research Site, George Town
  - Research Site, Johor Bahru
  - Research Site, Kuantan
  - Research Site, Kuching
- Research Site, Szczecin, Poland
- South Korea (5):
  - Research Site, Cheongju-si
  - Research Site, Donggu
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Research Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for individual participant data (IPD), but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home